CLINICAL TRIAL: NCT03907839
Title: Effects of Cognitive Training Combined With Pulmonary Rehabilitation on Exercise Tolerance and Cognitive Functions in COPD Patients: a Randomized Controlled Trial
Brief Title: Effects of Combined Cognitive Rehabilitation in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Imen Sanaa, PhD, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: pulmonary rehabilitation
Record Dates: First submitted 2019-04-03; First posted 2019-04-09 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-04

CONDITIONS: COPD
Keywords: COPD; cognitive training; cognitive impairment; P300 test; MOCA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction | interventions — Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance Training (ET) (Active Comparator): endurance training for control group
  Interventions: Other: clinical trials
- ET+cognitive training(CT) (Experimental): endurance training added to cognitive training for exprimental COPD group
  Interventions: Other: clinical trials

INTERVENTIONS:
Other: clinical trials — examined two type of training on cognitive parameters for COPD patients

SUMMARY:
This study was to examine the effect of endurance training combined with cognitive training in patients with COPD. The intervention group underwent Cognitive Training added to Endurance Training and the control group underwent only Endurance Training.

DETAILED DESCRIPTION:
Pulmonary rehabilitation is an essential part of the management of COPD. Although various methods and therapies of PR have been used in COPD patients. Furthermore, the Cognitive Training has been performed people with mild cognitive impairments.

Therefore, the combination of endurance training and cognitive tarining could be another alternative to improve the exercise tolerance and cognitive function in patients with COPD. It may also be useful for clinicians interested in designing new rehabilitation therapies. The aim of the study was to analyze the effect of CT combined with ET on exercise tolerance and cognitive functions in COPD patient.

ELIGIBILITY:
Inclusion Criteria:

* clinically stable COPD diagnosed by pulmonary function testing (2) absence of heart diseases, severe psychiatric, neurologic or musculoskeletal conditions and /or instable cardiovascular diseases. (3) Absence of medication influencing cognition (4) without history of brain injury, history of stroke or history of alcoholism.

Exclusion Criteria:

* smoking COPD
* heart diseases
* instable cardiovascular diseases

Ages: 60 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | 1 day
  The patients are instructed to cover the maximal distance in 6 min.Dyspnea was measured using Borg scale before the start of 6MWT and at the end of the test. Portable Spiropalm COSMED recorded heart rate (HR) and oxygen saturation (SpO2) continuously throughout the 6MWT. At the end of the 6MWT, the total covered distance was recorded.
Montreal cognitive assessment test | 1 day
  The test, scored on a scale of 0-30 points, is designed to identify cognitive impairment by assessing multiple cognitive domains.
  MOCA scores between 26 and 30 are consid¬ered normal, while scores < 26 indicate cognitive impairment
P300 test | 2 days
  The electroencephalogram signals were recorded with Fz, Cz, and Pz, electrodes. The P3b and P3a components were identified as the largest positive deflections between 250 ms and 500 ms, respectively, in the target and novel responses. Scalp electrode activity was measured at all electrode sites of which Fz, Cz, and Pz were analyzed. Fz, Cz, and Pz were chosen for analyses because ERPs responses are largest on the midline locations.

REFERENCES:
- [Background] Cleutjens FA, Janssen DJ, Ponds RW, Dijkstra JB, Wouters EF. COgnitive-pulmonary disease. Biomed Res Int. 2014;2014:697825. doi: 10.1155/2014/697825. Epub 2014 Mar 16. PMID 24738069
- [Background] Dodd JW, Charlton RA, van den Broek MD, Jones PW. Cognitive dysfunction in patients hospitalized with acute exacerbation of COPD. Chest. 2013 Jul;144(1):119-127. doi: 10.1378/chest.12-2099. PMID 23349026
- [Background] Bersani FS, Minichino A, Fattapposta F, Bernabei L, Spagnoli F, Mannarelli D, Francesconi M, Pauletti C, Corrado A, Vergnani L, Taddei I, Biondi M, Delle Chiaie R. Prefrontocerebellar transcranial direct current stimulation increases amplitude and decreases latency of P3b component in patients with euthymic bipolar disorder. Neuropsychiatr Dis Treat. 2015 Nov 19;11:2913-7. doi: 10.2147/NDT.S91625. eCollection 2015. PMID 26640377
- [Background] Kirkil G, Tug T, Ozel E, Bulut S, Tekatas A, Muz MH. The evaluation of cognitive functions with P300 test for chronic obstructive pulmonary disease patients in attack and stable period. Clin Neurol Neurosurg. 2007 Sep;109(7):553-60. doi: 10.1016/j.clineuro.2007.03.013. Epub 2007 May 29. PMID 17532116